CLINICAL TRIAL: NCT03371121
Title: Valutazione Dell'Epidemiologia e Dei Risultati Radiografici e Clinici Nel Trattamento Artroscopico Delle Lesioni Osteocondrali Dell'Astragalo Con Tecnica AMIC
Brief Title: Clinical and Radiographic Outcomes After AMIC Treatment for Talus Osteochondral Lesion Trattamento Artroscopico Delle Lesioni Osteocondrali Dell'Astragalo Con Tecnica AMIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMIC
Record Dates: First submitted 2017-12-07; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Talar Osteochondral Defect of Ankle; Pain; Arthroscopy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chondro-gide - Geistlich (Other): Arthroscopic use of chondro-gide to treat symptomatic osteochondral talar lesion
  Interventions: Other: AT-AMIC (arthroscopic talus autologous matrix induced chondrogenesis)

INTERVENTIONS:
Other: AT-AMIC (arthroscopic talus autologous matrix induced chondrogenesis) — to fill arthroscopically osteochondral talar lesion

SUMMARY:
Aim of the study is to evaluate clinical and radiographic outcomes in patients undergone all-arthroscopic autologous matrix induced chondrogenesis for symptomatic osteochondral talar lesions

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* males and females
* patients underwent arthroscopic cartilage reconstruction surgery with AMIC technique for osteochondral lesions of the talus

Exclusion Criteria:

* age <18 years at the time of surgery
* patients with previous surgery on the affected ankle

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2016-04-26 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Radiologic reduction of the lesion | 5 years
  A reduction of at least 30% of the lesion is to be expected

CONTACTS AND LOCATIONS:
Overall Officials: Federico G Usuelli, MD, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- Federico Usuelli, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided